CLINICAL TRIAL: NCT03367780
Title: Determining the Dose-Effect Relation of Salivary Gland Irradiation and Cell Loss With PSMA PET
Brief Title: Dose-Effect Relation of Salivary Gland Irradiation
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: N17DSI
Record Dates: First submitted 2017-11-20; First posted 2017-12-11 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-04

CONDITIONS: HNSCC
Keywords: Head-neck tumours; Radiotherapy; Salivary gland toxicity; PSMA PET/CT
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RT with curative intent for HNSCC: several schemes for radical (chemo)radiotherapy, administered in 30-35 fractions over 6-7 weeks
  Interventions: Device: PSMA PET/CT-scan

INTERVENTIONS:
Device: PSMA PET/CT-scan — PSMA PET is a new diagnostic instrument which can visualize the presence of vital acinar cells in salivary gland locations throughout the head and neck, with a sensitive and quantitative signal.

SUMMARY:
Optimization of radiotherapy to reduce xerostomia is difficult, because many gland locations cannot be seen with current imaging modalities and biological dose-effect are currently insufficiently understood. PSMA PET is a new diagnostic instrument which can visualize the presence of vital acinar cells in salivary gland locations throughout the head and neck, with a sensitive and quantitative signal. A reduction of PSMA accumulation in salivary glands is thought to correlate with loss of vital acinar cells. The PET images can be correlated with radiotherapy dose distributions in gland-based or voxel-based evaluations. This makes PSMA PET a suitable instrument to derive the radiobiological dose-effect relations that are required to develop better and gland-specific dose constraints for radiotherapy. The results of this study can contribute to lower toxicity and better quality of life in patients treated with high-dose radiotherapy in the head and neck.

DETAILED DESCRIPTION:
Primary objective of this prospective observational study is to determine the gland-based dose-effect relation between conventionally fractionated radiotherapy (RT) and long-term loss of acinar cells, per salivary gland type. The study population consists of a maximum of 20 patients with HNSCC referred for high-dose (CC)RT. There is no therapeutic intervention. Diagnostic intervention is PSMA PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* HNSCC of the head-neck area, cTx-4 N0-3 M0
* Accepted for EBRT in a conventionally fractionated schedule of 6-7 weeks.

Exclusion Criteria:

* Age <18y
* Pregnancy or lactation
* Participation in conflicting studies, e.g. with non-standard treatment and/or imaging
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven mucosal squamous cell carcinoma in the head-neck area who are referred for high dose EBRT based on current clinical criteria. AVL currently treats multiple new patients per week, and with an inclusion rate of 50% this observational study can complete inclusion well within one year. The study will close after 6 months of follow-up of the last included patient, for an expected total study duration of 1.5 years.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
the mean received radiation dose to salivary glands (Dmean), and the total uptake of PSMA in salivary glands (SUVtotal) and its relative reduction after radiotherapy (ΔSUVtotal-6). | 6 months
  Dmean and ΔSUVtotal-6 are correlated to determine the dose-effect relation.

SECONDARY OUTCOMES:
ΔSUV | 1 month
the clinical evaluation of a dry mouth | before treatment, once during 7 weeks of treatment and follow up 6 months after
  according to the C30+HN35 QoL
the clinical evaluation of a dry mouth | before treatment, once a week during 7 weeks of treatment and follow up 6 months after
  Groningen questionnaires
voxel-based ΔSUV | 7 weeks of treatment, follow-up 1 and 6 months
Voxel-based received radiation dose | 7 weeks of treatment, 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wouter V Vogel, MD,PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (3):
- Netherlands (3):
  - The Netherlands Cancer Institute- Antoni van Leeuwenhoek (NKI-AVL), Amsterdam, North Holland
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No